CLINICAL TRIAL: NCT06815562
Title: Placement Success Predictor: Using Site-Customized Machine Learning Models to Predict the Best Level of Care Placement for Each Child's Behavioral Health Needs
Brief Title: Predict the Best Level of Care Placement for Each Child's Behavioral Health Needs - Efficacy Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Outcome Referrals, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); State of Iowa Department of Health and Human Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R44MH125486-02A1-Aim 2A; 2R44MH125486-02A1 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Adolescent Well-Being; Mental Health Wellness

STUDY DESIGN:
Intervention Model Description: Efficacy (randomized clinical trial) study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Access to PSP site-specific placement prediction scores for that youth (Experimental): The PSP system will provide site-specific placement success prediction scores [i.e., client's likelihood of success per placement based on machine learning models] for each youth randomized to this condition in the efficacy study.
  Interventions: Other: Clinical team access to Placement Success Predictor (PSP) results
- No PSP site-specific placement prediction scores for that youth (No Intervention)

INTERVENTIONS:
Other: Clinical team access to Placement Success Predictor (PSP) results — PSP is a machine-learning based clinical decision support tool that is designed to assist clinical team members in making placement decisions for youth.
  Arms: Access to PSP site-specific placement prediction scores for that youth

SUMMARY:
The purpose of this randomized clinical trial is to test the efficacy of a new clinical decision support tool, Placement Success Predictor (PSP). PSP will provide placement-specific predictions about the likelihood of a youth having a good outcome in each placement type using machine learning algorithms.

The primary hypothesis is that if clinical team members have access to PSP results for youth in the experimental group, these youth will have better outcomes at the 3-month follow-up compared to youth in the control group.

DETAILED DESCRIPTION:
In 2017, a total of 669,799 children were confirmed victims of maltreatment in the United States; of the 442,733 children in foster care, 34% have been in more than one placement and 11% are in a group home or institution. Stakes are extremely high for making the best out-of-home placement choice per child because some placement types and multiple placements are associated with poor outcomes. In the past few years, legislation has been created to guide placement decisions for children. Federal law 42 U.S. Code 675 requires that children in the care of the state are placed "in a safe setting that is the least restrictive (most family like)." In addition, the Family First Prevention Services Act signed into law by the U.S. Congress in 2018 includes measures to reduce the number of children in long-term residential settings. This study is an effort to develop and test a science-based clinical decision support tool using behavioral health data collected through standard clinical practice.

A randomized controlled trial (RCT) design will be used to assess efficacy of clinical team access to Placement Success Predictor (PSP) on child welfare clients' well-being outcomes and healthcare costs.

Sample. Clients at the State of Iowa Department of Health and Human Services (Iowa HHS) are the sample for this efficacy study.

Randomization. The outcome of a single coin toss was applied to an undisclosed algorithm for the client's record number to determine who gets assigned to the experimental group (i.e., client has PSP results).

Methods. The Treatment Outcome Package (TOP), a behavioral health assessment, is a standard part of care delivered in Iowa and its completion is required by the state. Iowa HHS clinical teams will be provided PSP results for clients in the experimental condition. A request for a waiver of consent for this study was approved by the WCG IRB.

ELIGIBILITY:
Inclusion Criteria:

* Completed TOP CS assessment

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference on average z-scores across raters within two weeks on the Clinical Scale of the Treatment Outcome Package (TOP-CS) between a) the beginning of the study (between February and October 2025) and b) approximately 3 months later. | At baseline and in 3 months
  TOP is a comprehensive well-being assessment that is used in behavioral health and child welfare settings. The Child TOP Clinical Scale (TOP-CS) is a 58-item scale for children (ages 3 - 18) that assesses 13 domains. The Adolescent TOP Clinical Scale (TOP-CS) is a 48-item scale for adolescents (ages 11 - 21) that assesses 12 domains. TOP-CS assesses the client's past 2-week experience on domains including Depression, Violence, and Suicidality (scores are risk-adjusted for case mix variables assessed via 37 items on the companion TOP-Case Mix form regarding stressful life events, comorbidity). Participants answer "All" to "None of the Time" for each item on a 6-point Likert scale. The z-scores (standard deviation units relative to the general population mean for each domain) will be averaged together to create one summary score. Higher scores suggest higher severity/lower behavioral well-being.

SECONDARY OUTCOMES:
Total cost of treatment | 3 months
  Estimated treatment cost per placement per participant will be assessed by calculating the number of days in treatment times cost per day
Mean difference on average z-scores across raters within two weeks on the TOP-CS between a) the PREDICTED [i.e., risk-adjusted] scores at beginning of the study and b) the ACTUAL follow up scores approximately 3 months later. | At baseline and in 3 months
  See Outcome description 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Outcome Referrals, Inc., Framingham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trudeau KJ, Yang J, Di J, Lu Y, Kraus DR. Predicting Successful Placements for Youth in Child Welfare with Machine Learning. Child Youth Serv Rev. 2023 Oct;153:107117. doi: 10.1016/j.childyouth.2023.107117. Epub 2023 Aug 4. PMID 37841819
- [Background] Kraus DR, Seligman DA, Jordan JR. Validation of a behavioral health treatment outcome and assessment tool designed for naturalistic settings: The Treatment Outcome Package. J Clin Psychol. 2005 Mar;61(3):285-314. doi: 10.1002/jclp.20084. PMID 15546147